CLINICAL TRIAL: NCT00181649
Title: Recombinant Human Prolactin for Lactation Induction in Adoptive Mothers
Brief Title: Recombinant Human Prolactin for Lactation Induction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not able to recruit any subjects.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Corrine Welt, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003P001209-2
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Lactation
Keywords: Lactation; Breastfeeding; Adoptive mothers; Prolactin; Relative lactation insufficiency
MeSH Terms: conditions — Breast Feeding

ARMS (1):
- Recombinant human prolactin (Experimental)
  Interventions: Drug: Recombinant human prolactin

INTERVENTIONS:
Drug: Recombinant human prolactin

SUMMARY:
The purpose of the study is to assess the safety and determine the effects of the hormone prolactin on lactation (breast milk production).

DETAILED DESCRIPTION:
Subjects will participate in a randomized, double-blind, placebo-controlled, crossover trial comparing breast pumping, alone, to breast pumping and r-hPRL. Subjects will have one week of instruction with the breast pump alone. Subsequently, subjects will receive 2 weeks of r-hPRL or placebo followed by 2 weeks of the alternate treatment.

Week 1: Study day 1, a baseline prolactin level will be obtained and subjects will be taught to use an electrical, hospital grade breast pump by a designated lactation consultant. Subjects will pump for 10 minutes at each breast. The total volume of milk will be recorded in a diary throughout the study. Prolactin levels will be obtained every 10 minutes for 60 minutes after pumping begins, then every 30 minutes for a total of 3 hours. Subjects will pump 3 times per day increasing to 8 times per day by the end of the first week and will continue this regimen throughout the study.

Week 2: One week after the initial visit, subjects will return to the GCRC for re-evaluation of the pumping technique and the first dose of medication. Subjects will pump for 10 minutes at each breast as on day 1 and prolactin levels will be obtained every 10 minutes for 60 minutes, then every 30 minutes for a total of 3 hours. At 3 hours, r-hPRL 60 mg/kg or placebo will be administered SC. Blood will be drawn every 10 minutes for 60 minutes, every 30 minutes for 2 hours, then at 4, 6 and 8 hours to obtain a peak prolactin level. Vital signs will be monitored every 15 minutes for the first hour, then every 2 hours for a total of 8 hours. Subjects will pump both breasts every 3 hours, starting after the r-hPRL or placebo injection. Subjects will be taught to give themselves SC injections and will administer their second dose of SC r-hPRL or placebo 12 hours after the first dose. Subjects will continue SC r-hPRL or placebo administration every 12 hours for the next 14 days. They will continue to pump daily, approximately every 3 hours, with a 5 hour break in the night to sleep. Subjects will be asked to refrigerate all milk and bring it in to GCRC visits for prolactin levels.

Subjects will return weekly for 4 additional visits (weeks 3, 4, 5, 6). At the weekly visits, blood will be drawn at baseline for a prolactin level and r-hPRL or placebo will be administered. Blood will then be drawn every 10 minutes for 60 minutes, then every 30 minutes for 2 hours, then every 2 hours for a total of 8 hours after the injection. Vital signs will be monitored as described above. At the week 4 visit, subjects will be switched to the alternate treatment for weeks 4 and 5. Subjects will be seen 14 days after their final injection. A baseline prolactin level will be drawn, then milk will be pumped, as previously. Blood will be drawn every 10 minutes for 60 minutes, then every 30 minutes for a total of 3 hours. A 1 cc sample of the milk will also be obtained 14 days after the final injection for analysis of composition. All side effects of r-hPRL will be recorded throughout the study. All milk obtained during the study will be stored and the milk composition will be determined before it is used. Infants receiving milk produced during the study will initially be monitored in the GCRC under the supervision of a neonatologist.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-postpartum women, aged 18-45 years, who desire to lactate for their adoptive children
* Normal thyroid-stimulating hormone (TSH) and prolactin level
* Normal adrenal gland function or taking physiological glucocorticoid replacement
* No medical illnesses that contraindicate breastfeeding
* HIV negative
* Normal breast development

Exclusion Criteria:

* Use of medications known to increase prolactin
* Anatomical breast abnormalities
* Previous mammoplasty or breast augmentation
* Current use of hormonal contraception
* Allergies to mannitol
* Medications contraindicated for breastfeeding mothers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Breast milk production | 28 days

SECONDARY OUTCOMES:
Breast milk volume | 28 days
Breast milk prolactin levels and content | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Corrine K Welt, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Powe CE, Puopolo KM, Newburg DS, Lonnerdal B, Chen C, Allen M, Merewood A, Worden S, Welt CK. Effects of recombinant human prolactin on breast milk composition. Pediatrics. 2011 Feb;127(2):e359-66. doi: 10.1542/peds.2010-1627. Epub 2011 Jan 24. PMID 21262884
- [Result] Powe CE, Allen M, Puopolo KM, Merewood A, Worden S, Johnson LC, Fleischman A, Welt CK. Recombinant human prolactin for the treatment of lactation insufficiency. Clin Endocrinol (Oxf). 2010 Nov;73(5):645-53. doi: 10.1111/j.1365-2265.2010.03850.x. PMID 20718766